CLINICAL TRIAL: NCT01115127
Title: Myo-inositol and Melatonin in Menopausal Transition. A Prospective, Randomized Trial
Brief Title: Myo-inositol and Melatonin in Pre-menopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, Myo-inositol and melatonin in menopausal transition., University of Messina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Myo-Mela-2010
Record Dates: First submitted 2010-04-22; First posted 2010-05-04 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Pre-menopausal Irregular Cycles and Bleedings
Keywords: pre-menopause; melatonin; myo-inositol
MeSH Terms: interventions — Melatonin; Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- myo-inositol (Active Comparator): 30 subjects will take 2 tablets per day containing 2 grams of myo-inositol, for 6 months.
  Interventions: Dietary Supplement: myo-inositol
- melatonin (Active Comparator): 30 subjects will take 1 tablet per day (at night-time) containing 3 grams of melatonin for 6 months
  Interventions: Dietary Supplement: melatonin
- melatonin plus myo-inositol (Active Comparator): 30 subjects will take 2 grams per day of myo-inositol and 3 grams of melatonin at night-time for 6 months
  Interventions: Dietary Supplement: melatonin plus myo-inositol

INTERVENTIONS:
Dietary Supplement: melatonin — 30 subjects will take 1 tablet per day (at night-time) containing 3 grams of melatonin for 6 months
  Arms: melatonin
Dietary Supplement: myo-inositol — 30 subjects will take 2 tablets per day containing 2 grams of myo-inositol, for 6 months.
  Arms: myo-inositol
Dietary Supplement: melatonin plus myo-inositol — 30 subjects will take 2 grams per day of myo-inositol and 3 grams of melatonin at night-time for 6 months
  Arms: melatonin plus myo-inositol

SUMMARY:
The purpose of this study is to determine whether myo-inositol and melatonin, or myo-inositol alone, or melatonin alone, are effective in normalizing irregular bleeding and anovulatory cycles in pre-menopausal women.

DETAILED DESCRIPTION:
Melatonin has produced a remarkable significant improvement of thyroid function, positive changes of gonadotropins towards reduced levels, and in some women a re-acquisition of normal menstrual cycle. Furthermore, an abrogation of menopause-related depression, amelioration of hot-flashes and improvement of quality and duration of sleep has been reported.

Myo-inositol is involved in several aspects of human reproduction. Elevated concentrations of myo-inositol in human follicular fluids appear to play a positive function in follicular maturity and provide a marker of good quality oocytes. Nevertheless its positive role in PCOS women is a consequence of a defect in the insulin signalling pathway (inositol-containing phosphoglycan mediators) that seems to be primarily implicated in the pathogenesis of insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* all pre-menopausal women with irregular cycles and bleedings

Exclusion Criteria:

* pre-menopausal women who take hormonal drugs

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Normalizing irregular bleeding and anovulatory cycles in pre-menopausal women. | 12 months

SECONDARY OUTCOMES:
Serum assays of thyroid hormones. | 12 months
Assays of gonadotropins and estradiol serum levels | 12 months
Evaluation of metabolic markers (insulin, glucose, total cholesterol, HDL-cholesterol, triglycerides). | 12 months
Variation of blood pressure. | 12 months
Variation of mood, hot flashes, quality of sleep. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, MD, Principal Investigator — University of Messina
Locations (1):
- University Hospital, Messina, Italy